CLINICAL TRIAL: NCT01203085
Title: Development and Validation of CMT Pediatric Scale for Children With Charcot Marie Tooth
Brief Title: Development of Charcot Marie Tooth Disease (CMT) Pediatric Scale for Children With CMT
Acronym: INC-6603
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Muscular Dystrophy Association (Other); University of Rochester (Other); Children's Hospital of Philadelphia (Other); University College London Hospitals (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Sydney Children's Hospitals Network (Other); Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Michael Shy, Professor, University of Iowa
Other Study IDs: INC-6603; 1U54NS065712-01 (NIH)
Record Dates: First submitted 2010-08-09; First posted 2010-09-16 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Charcot Marie Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric patients: All patients 21 years of age and under who are enrolled in the 6601 study and have undergone the pediatric scale tests.

SUMMARY:
The primary goal of this project is to develop and test a Charcot Marie Tooth disease (CMT) Pediatric Scale for use in evaluation in natural history CMT study.

DETAILED DESCRIPTION:
This project is to develop a new CMT Pediatric Scale (CMTPeds) for Children with CMT. Although there is a validated score (the CMTNS) which measures disease severity for CMT, it is not always applicable to children due to their limited ability to relay information about their symptoms. The CMTPeds scale is being developed and validated in order to measure disease severity in children and have outcome measures available for future clinical trials. Children (defined as 21 and under) being evaluated will be asked to perform functional tasks such as using stairs, walking in a hallway, and performing hand function tests. This information will be used to validate the CMTPeds score. It is important to have validated instruments to measure disease severity in childhood so these can be used with clinical treatment trials are available.

ELIGIBILITY:
Inclusion Criteria:

All patients MUST be seen in person at one of the participating centers for enrollment in this study.

* Children (< 21 years of age)
* Known or probable inherited neuropathies classified as CMT1, CMT2, or CMT4

Exclusion Criteria:

* Known diagnoses of acquired neuropathy including toxic (e. g. medication related neuropathies); metabolic (e.g. diabetic), immune mediated or inflammatory [acute inflammatory demyelinating polyradiculoneuropathy (AIDP) or chronic inflammatory demyelinating polyneuropathy (CIDP)] polyneuropathies; neuropathy related to leukodystrophy, congenital muscular dystrophy; and patients with severe general medical conditions.
* Entirely normal conduction velocities of upper and lower limbs as this suggests that the subject may not have a neuropathy.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are 21 years of age and under who are also enrolled in the 6601 study and have performed all tasks to complete the CMT Peds Scale will be recruited for participation. Participation entails allow the information collected in the 6601 study be used for validation in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
CMT Peds Scale Part 1: Symptoms | 1 year
  The CMT Peds Scale Symptoms include foot and hand symptoms.
CMT Peds Score Part 2: Foot and Ankle Involvement | 1 year
  Foot and ankle involvement includes foot posture index, range of ankle dorsiflexion, foot drop present/absent, and whether or not difficulty heel/toe walking.
CMT Peds Scale Part 3: Hand dexterity | 1 year
  Hand dexterity involves hand dexterity testing and the nine-hole peg test.
CMT Peds Scale Part 4: Hand strength | 1 year
  Hand strength includes grip strength, thumb-index pinch, and three point pinch.
CMT Peds Scale Part 5: Foot Strength | 1 year
  Foot strength includes the strength of plantar- and dorsi-flexion, eversion, and inversion.
CMT Peds Score Part 6: Sensation | 1 year
  Sensation includes pinprick and vibration sensations.
CMT Peds Scale Part 7: Balance | 1 year
  Balance is assessed by the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition (BOT-2).
CMT Peds Scale Part 8: Motor Function | 1 year
  Motor function assessment includes long jump, 10 meter run/walk, stair climb, stair descend, and 6 minute walk test.

SECONDARY OUTCOMES:
Evaluate CMT Pediatric Scale (CMT Peds Scale) in CMT natural history study | 6 months to 1 year
  The sections of the CMT Peds Scale which are found to be clinically/functionally useful after one year of analysis will be carried forward for all pediatric patients every 6 months to one year.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shy, MD, Principal Investigator — University of Iowa
Locations (14):
- United States (9):
  - Stanford University, Palo Alto, California
  - University of Connecticut/Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Children's Hospital of Westmead, Sydney, New South Wales, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- C. Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- United Kingdom (2):
  - National Hospital of Neurology and Neurosurgery, London, England
  - Dubowitz Neuromuscular Centre, London, UK

IPD SHARING:
Plan to Share IPD: Yes
De-identified RDCRN data is submitted to an ORDR-designated repository. For the current grant cycle, that repository has been dbGaP.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: (For Observational/Longitudinal/Natural History/Epidemiology studies): For the current grant cycle, available data will be released to the repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first.
Access Criteria: For the current grant cycle, once de-identified data is posted on dbGaP, a summary of the study is posted and individual participant data is accessed via a request through dbGaP.
URL: https://www.ncbi.nlm.nih.gov/projects/gap/cgi-bin/study.cgi?study_id=phs001553.v1.p1

REFERENCES:
- See also: Inherited Neuropathy Consortium Website — https://www1.rarediseasesnetwork.org/cms/inc